CLINICAL TRIAL: NCT04172350
Title: Developing and Examining Preliminary Effects of An Innovative Care-improvement Smartphone-based Perioperative Solution for Women Undergoing Breast Cancer Surgery (iCareBreast): A Pilot Randomized Controlled Trial
Brief Title: An Innovative Care-improvement Smartphone-based Perioperative Solution for Women Undergoing Breast Cancer Surgery
Acronym: iCareBreast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HE Hong-Gu (Other)
Collaborators: KK Women's and Children's Hospital (Other Government); Buddy Healthcare Ltd OY (Unknown)
Responsible Party: Sponsor-Investigator, HE Hong-Gu, Associate Professor, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019/2632
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer Female; Surgery
Keywords: women; breast cancer; surgery; perioperative care; self-efficacy; randomised controlled trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A two-group pre- and post-test randomized controlled trial will be conducted. A total of 112 eligible women who are diagnosed with breast cancer and are required for breast surgery will be recruited from the Breast Department in a public tertiary hospital in Singapore. Participants will be randomly allocated to either the intervention group (receiving routine care provided by the hospital plus iCareBreast) or the control group (only receiving routine care provided by the hospital) using a block randomisation.
Who Masked: Outcomes Assessor
Masking Description: The principal investigator will generate the randomisation number and randomisation sequences according to the block randomisation method. The randomly generated sequences would be used for recruitment of the participants, who will be assigned in successive order according to the sequence. Opaque and sealed envelopes containing slips of paper indicate the randomly allocated group. One research assistant will recruit participants and conduct randomisation and another research assistant who is blind from the group allocation will collect post-test data. Through these carefully deliberated processes, randomization and allocation concealment will be ensured.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: iCareBreast plus routine care (Experimental): Participants in the intervention group will receive the routine care provided by the hospital (the same as the control group) plus the iCareBreast mobile app, which provides i) pre-surgery education and instructions; ii) post-surgery education, instructions, and recovery plan; iii) positive psychological support; and iv) social support. The total intervention period is 29 days (14 days before surgery, operation day, and 14 days after the surgery).
  Interventions: Other: iCareBreast; Other: Routine care
- Control group: Routine care (Active Comparator): Participants in the control group will only receive routine care provided by the attending Hospital. Participants being allocated to the control group may freely use the Internet to search for information regarding breast cancer but will not be granted to access the iCareBreast app.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: iCareBreast — The iCareBreast BuddyCare mobile app is an interactive surgery preparation and recovery app for patients. It is a patient-centric care coordination and patient engagement mobile app that supports patients' perioperative journey. The app provides day-to-day information throughout the perioperative journey to patients from 2 weeks before surgery to 2 weeks after the surgery. Meanwhile the healthcare professional can monitor patients' use of the app. That is, the iCareBreast App provides patients with all the information about the surgery-related procedure and treatment via an efficient, user-friendly and interactive timeline. Patients will receive pop-up reminders daily for them to use the app. The objective of this app is to allow each patient to focus on caring for herself as a patient.
  Arms: Intervention group: iCareBreast plus routine care
Other: Routine care — Routine care provided by the hospital includes general information regarding pre-operation preparation and post-operative care (e.g. wound care, pain management and physiotherapy).

SUMMARY:
This study aims to develop a mobile app-based periopeartive intervnetion for women undergoing breast cancer surgery and examine the effectiveness of the program on participants' health outcomes of self-efficacy, anxiety and depression, pain and fatigue, quality of life, and satisfaction with perioperative care. This study also aims to explore the perceptions of participants on strengths and weaknesses of using the app.

DETAILED DESCRIPTION:
Background: Breast cancer is the most common cancer in women worldwide and Singapore. In addition to the disease itself, undergoing surgery is also a stressful event for patients. Many of them have physical and psychosocial challenges. A variety of psychosocial interventions have been developed to improve patients'/survivors' health outcomes with some intervention using mobile technology. However, there is no any smart-phone based solution that have developed a comprehensive perioperative solution for this group of patients.

Aim: This study aims to (1) develop an Innovative Care-improvement Smartphone-based Perioperative Solution for Women Undergoing Breast Cancer Surgery (iCareBreast); (2) examine the effectiveness of the iCareBreast on participants' health outcomes of self-efficacy (primary outcome), anxiety and depression, pain and fatigue, quality of life, and satisfaction with perioperative care; and (3) explore the perceptions of participants on strengths and weaknesses of iCareBreast.

Research Questions:

* Do the participants receiving routine care plus the iCareBreast report higher level of self-efficacy when compared to those receiving routine care alone?
* Do the participants receiving routine care plus the iCareBreast report lower levels of anxiety and depression when compared to those receiving routine care alone?
* Do the participants receiving routine care plus the iCareBreast report lower levels of postoperative pain and fatigue when compared to those in the control group?
* Do the participants receiving routine care plus the iCareBreast report higher level of quality of life when compared to those receiving routine care alone?
* Do the participants receiving routine care plus the iCareBreast report higher level of satisfaction with perioperative care when compared to those receiving routine care alone?
* What are the perceptions of participants on strengths and weaknesses of iCareBreast?

Hypothesis As compared to the participants in the control group, those in the intervention group who receive routine care plus the iCareBreast will report a

* higher level of self-efficacy,
* lower levels of anxiety and depression,
* lower levels of pain and fatigue,
* higher level of quality of life, and
* higher level of satisfaction with perioperative care.

Methods: A two-group pre- and post-test randomized controlled trial will be conducted. A total of 112 eligible women who are diagnosed with breast cancer and are required for breast surgery will be recruited from the Breast Department in a public tertiary hospital in Singapore. Participants will be randomly allocated to either the intervention group (receiving routine care provided by the hospital plus iCareBreast) or the control group (only receiving routine care provided by the hospital). Outcomes of self-efficacy, anxiety and depression, pain and fatigue, quality of life, and satisfaction with perioperative care will be measured by relevant valid and reliable instruments at two time-points (baseline and post-test). Around 15 participants in the intervention group will be invited to participate in semi-structured interviews to explore their opinions on the iCareBreast. Quantitative data will be analyzed by SPSS and qualitative data will be analyzed by using content analysis.

Significance of the study: This study will develop the iCareBreast, which will provide a platform for women undergoing breast cancer surgery to receive education about the disease, physical, psychological and social support as well as to enable interactions between health care workers and patients. This study will generate the preliminary effects of the iCareBreast to improve the aforementioned health outcomes of participants, which will be used to guide the change of future clinical practice to improve patient care. Mobile health holds promise as a low-cost communication tool for enhancing patient engagement and allowing healthcare providers to monitor recovery progress. This study will also inform the need for further studies for the implementation of similar solution for patients with other surgical needs.

ELIGIBILITY:
Inclusion Criteria:

* are the age of 21 years old and above at the point of recruitment;
* are diagnosed with breast cancer;
* will undergo breast cancer surgery (mastectomy or wide excision);
* can speak, read and write in English; and
* has access to smart phone.

Exclusion Criteria:

* been suffering from psychiatric illness or impaired cognitive function;
* alcohol or substance abuse within the previous year;
* anxiety disorder and other mood disorder as identified from their medical records; and
* been in the bereavement period in the last 6 months.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Participant's self-efficacy | Participant's self-efficacy will be assessed at baseline (about 2 weeks before surgery) and assessing changes between baseline and 2 weeks after surgery.
  Participant's self-efficacy level will be measured using the 10-item General Self-Efficacy (GSE) Scale. The total score for GSE is tabulated by the sum of all scores of each component. The scoring system ranges between 10 and 40. The higher the score achieved, the higher the level of self-efficacy (Schwarzer & Jerusalem, 1995).

SECONDARY OUTCOMES:
Participant's anxiety and depression | Participant's anxiety and depression will be assessed at baseline (about 2 weeks before surgery) and assessing changes between baseline and 2 weeks after surgery.
  Participant's anxiety and depression levels will be measured using the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 items: 7 items measuring depression and the other 7 items measuring anxiety. The response ranges from 0 (no problem) to 3 (high level of problem). The total score ranged from 0 to 21 with the higher score indicating more anxiety or depression.
Participant's pain and fatigue | Participant's pain and fatigue will be assessed at baseline (about 2 weeks before surgery) and assessing changes between baseline and 2 weeks after surgery.
  Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) will be used to measure participant's pain and fatigue level in this study. The MFSI-SF consists of 30 items. Respondents indicate the extent to which they have experienced each symptom during the preceding one-week period (0 = not at all; 4 = extremely). Ratings are summed to obtain scores for 5 subscales (general fatigue, physical fatigue, emotional fatigue, mental fatigue, and vigor) with the higher score indicating worse symptom.
Participant's quality of life | Participant's quality of life will be assessed at baseline (about 2 weeks before surgery) and assessing changes between baseline and 2 weeks after surgery.
  Participant's quality of life will be measured by the European Organization for Research and Treatment-QOL questionnaire and breast cancer specific module (EORTC QLQ-BR23). The format uses Likert scales, with scoring from 1 ('not at all') to 4 ('very much'). The EORTC QLQ-BR23 is a breast-specific module that comprises of 23 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss. The scoring of the EORTC QLQ-BR23 was performed according to the EORTC scoring manual. All scores were linearly transformed to a 0 to 100 scale with a higher functional score representing a more healthy level of functioning, while a higher symptom score represents a worse symptom/problem.
Satisfaction with perioperative care | Participant's satisfaction with perioperative care will be assessed around 2 weeks after surgery.
  A 6-point Ordinal Descriptive Scale (ODS) for assessing patients' satisfaction with perioperative care from 1 (very dissatisfied) to 6 (very satisfied) will be used to assess patients' self-reported level of satisfaction with perioperative care they received.
Process evaluation interview | Semi-structured interviews will be conducted around 2 weeks after surgery.
  A semi-structured interview guide will be used to interview about 15 participants from the intervention group for their opinion on the strengths, weaknesses of the iCareBreast, as well as their suggestions for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Gu HE, PhD, Principal Investigator — National University of Singapore
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreu Vaillo Y, Murgui Perez S, Martinez Lopez P, Romero Retes R. Mini-Mental Adjustment to Cancer Scale: Construct validation in Spanish breast cancer patients. J Psychosom Res. 2018 Nov;114:38-44. doi: 10.1016/j.jpsychores.2018.09.004. Epub 2018 Sep 15. PMID 30314577
- [Background] Beck KR, Tan SM, Lum SS, Lim LE, Krishna LK. Validation of the emotion thermometers and hospital anxiety and depression scales in Singapore: Screening cancer patients for distress, anxiety and depression. Asia Pac J Clin Oncol. 2016 Jun;12(2):e241-9. doi: 10.1111/ajco.12180. Epub 2014 Mar 27. PMID 24673756
- [Background] Bener A, Alsulaiman R, Doodson L, El Ayoubi HR. An assessment of reliability and validity of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 among breast cancer patients in Qatar. J Family Med Prim Care. 2017 Oct-Dec;6(4):824-831. doi: 10.4103/jfmpc.jfmpc_17_17. PMID 29564271
- [Background] Boesen EH, Karlsen R, Christensen J, Paaschburg B, Nielsen D, Bloch IS, Christiansen B, Jacobsen K, Johansen C. Psychosocial group intervention for patients with primary breast cancer: a randomised trial. Eur J Cancer. 2011 Jun;47(9):1363-72. doi: 10.1016/j.ejca.2011.01.002. Epub 2011 Mar 31. PMID 21458989
- [Background] Bradley EH, Curry LA, Devers KJ. Qualitative data analysis for health services research: developing taxonomy, themes, and theory. Health Serv Res. 2007 Aug;42(4):1758-72. doi: 10.1111/j.1475-6773.2006.00684.x. PMID 17286625
- [Background] Brady L. My Journey With Triple Negative Breast Cancer. Plast Surg Nurs. 2015 Jul-Sep;35(3):137-44. doi: 10.1097/PSN.0000000000000107. No abstract available. PMID 26313679
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3(2), 77-101.
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Braybrooke JP, Mimoun S, Zarca D, Elia D, Pinder B, Lloyd AJ, Breheny K, Lomazzi M, Borisch B. Patients' experiences following breast cancer treatment: an exploratory survey of personal and work experiences of breast cancer patients from three European countries. Eur J Cancer Care (Engl). 2015 Sep;24(5):650-61. doi: 10.1111/ecc.12222. Epub 2014 Jul 23. PMID 25053521
- [Background] Broglio K. Randomization in Clinical Trials: Permuted Blocks and Stratification. JAMA. 2018 Jun 5;319(21):2223-2224. doi: 10.1001/jama.2018.6360. No abstract available. PMID 29872845
- [Background] Chan A, Lew C, Wang XJ, Ng T, Chae JW, Yeo HL, Shwe M, Gan YX. Psychometric properties and measurement equivalence of the Multidimensional Fatigue Syndrome Inventory- Short Form (MFSI-SF) amongst breast cancer and lymphoma patients in Singapore. Health Qual Life Outcomes. 2018 Jan 19;16(1):20. doi: 10.1186/s12955-018-0846-6. PMID 29351803
- [Background] Chaoul A, Milbury K, Spelman A, Basen-Engquist K, Hall MH, Wei Q, Shih YT, Arun B, Valero V, Perkins GH, Babiera GV, Wangyal T, Engle R, Harrison CA, Li Y, Cohen L. Randomized trial of Tibetan yoga in patients with breast cancer undergoing chemotherapy. Cancer. 2018 Jan 1;124(1):36-45. doi: 10.1002/cncr.30938. Epub 2017 Sep 20. PMID 28940301
- [Background] Chenail, R. J. (2011). How to conduct clinical qualitative research on the patient's experience. Qualitative Report, 16(4), 1173-1190.
- [Background] Cobo-Cuenca AI, Martin-Espinosa NM, Rodriguez-Borrego MA, Carmona-Torres JM. Determinants of satisfaction with life and self-esteem in women with breast cancer. Qual Life Res. 2019 Feb;28(2):379-387. doi: 10.1007/s11136-018-2017-y. Epub 2018 Oct 15. PMID 30324585
- [Background] Coyne IT. Sampling in qualitative research. Purposeful and theoretical sampling; merging or clear boundaries? J Adv Nurs. 1997 Sep;26(3):623-30. doi: 10.1046/j.1365-2648.1997.t01-25-00999.x. PMID 9378886
- [Background] Cramer H, Lange S, Klose P, Paul A, Dobos G. Yoga for breast cancer patients and survivors: a systematic review and meta-analysis. BMC Cancer. 2012 Sep 18;12:412. doi: 10.1186/1471-2407-12-412. PMID 22988934
- [Background] de Boer M, Zeiler K, Slatman J. Sharing lives, sharing bodies: partners negotiating breast cancer experiences. Med Health Care Philos. 2019 Jun;22(2):253-265. doi: 10.1007/s11019-018-9866-6. PMID 30191500
- [Background] Diekmann A, Heuser C, Ernstmann N, Geiser F, Gross SE, Midding E, Pfaff H, Ansmann L. How do breast cancer patients experience multidisciplinary tumor conferences? - A description from the patient perspective. Breast. 2019 Apr;44:66-72. doi: 10.1016/j.breast.2018.12.012. Epub 2019 Jan 4. PMID 30669033
- [Background] Droog E, Armstrong C, MacCurtain S. Supporting patients during their breast cancer journey: the informational role of clinical nurse specialists. Cancer Nurs. 2014 Nov-Dec;37(6):429-35. doi: 10.1097/NCC.0000000000000109. PMID 24406379
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Fillon M. Perioperative management may lead to less pain after breast cancer surgery. CA Cancer J Clin. 2019 Jan;69(1):5-6. doi: 10.3322/caac.21465. Epub 2018 Nov 26. No abstract available. PMID 30475405
- [Background] Gokal K, Wallis D, Ahmed S, Boiangiu I, Kancherla K, Munir F. Effects of a self-managed home-based walking intervention on psychosocial health outcomes for breast cancer patients receiving chemotherapy: a randomised controlled trial. Support Care Cancer. 2016 Mar;24(3):1139-66. doi: 10.1007/s00520-015-2884-5. Epub 2015 Aug 15. PMID 26275768
- [Background] Guarda Korelo RI, Siega J, Cordeiro Woloschen AC, Paula do Amaral M, Barao Dos Santos Ivanski M, Schleder JC, Fernandes LC. Brazilian Version of Cancer Fatigue Scale: Validation of the Brazilian Version of Cancer Fatigue Scale in Patients With Breast Cancer. J Pain Symptom Manage. 2019 Jun;57(6):1130-1136. doi: 10.1016/j.jpainsymman.2019.03.011. Epub 2019 Mar 21. PMID 30904416
- [Background] Guest, G., Bunce, A., & Johnson, L. (2006). How many interviews are enough? An experiment with data saturation and variability. Field Methods, 18(1), 59-82.
- [Background] Guilford, K., McKinley, E., & Turner, L. (2017). Breast cancer knowledge, beliefs, and screening behaviors of college women: Application of the health belief model. American Journal of Health Education, 48(4), 256-263. doi:10.1080/19325037.2017.1316694
- [Background] Hallowell N, Baylock B, Heiniger L, Butow PN, Patel D, Meiser B, Saunders C; kConFab Psychosocial Group on behalf of the kConFab Investigators; Price MA. Looking different, feeling different: women's reactions to risk-reducing breast and ovarian surgery. Fam Cancer. 2012 Jun;11(2):215-24. doi: 10.1007/s10689-011-9504-4. PMID 22198037
- [Background] Hauffman A, Alfonsson S, Mattsson S, Forslund M, Bill-Axelson A, Nygren P, Johansson B. The Development of a Nurse-Led Internet-Based Learning and Self-care Program for Cancer Patients With Symptoms of Anxiety and Depression-A Part of U-CARE. Cancer Nurs. 2017 Sep/Oct;40(5):E9-E16. doi: 10.1097/NCC.0000000000000402. PMID 27223884
- [Background] Heinze SB, Williams PD. Symptom alleviation and self-care among breast cancer survivors after treatment completion. Clin J Oncol Nurs. 2015 Jun;19(3):343-9. doi: 10.1188/15.CJON.343-349. PMID 26000584
- [Background] Higginbottom GM. Sampling issues in qualitative research. Nurse Res. 2004;12(1):7-19. doi: 10.7748/nr2004.07.12.1.7.c5927. PMID 15493211
- [Background] Ho RT, Potash JS, Fu W, Wong KP, Chan CL. Changes in breast cancer patients after psychosocial intervention as indicated in drawings. Psychooncology. 2010 Apr;19(4):353-60. doi: 10.1002/pon.1551. PMID 19358159
- [Background] Holloway, I., & Wheeler, S. (2002). Qualitative Research in Nursing (2nd edn). Oxford: Blackwell Science Ltd.
- [Background] Keilmann, L., Matthies, L., Simoes, E., Hartkopf, A. D., Sokolov, A. N., Walter, C. B., . . . Graf, J. (2019). Quality of life measurement in breast cancer patients: Reliability of an ePRO tool using EORTC QLQ-C30. European Journal of Obstetrics & Gynecology and Reproductive Biology, 234, e148-e149. doi:10.1016/j.ejogrb.2018.08.483
- [Background] Kim J, Lim S, Min YH, Shin YW, Lee B, Sohn G, Jung KH, Lee JH, Son BH, Ahn SH, Shin SY, Lee JW. Depression Screening Using Daily Mental-Health Ratings from a Smartphone Application for Breast Cancer Patients. J Med Internet Res. 2016 Aug 4;18(8):e216. doi: 10.2196/jmir.5598. PMID 27492880
- [Background] Kyranou M, Puntillo K, Dunn LB, Aouizerat BE, Paul SM, Cooper BA, Neuhaus J, West C, Dodd M, Miaskowski C. Predictors of initial levels and trajectories of anxiety in women before and for 6 months after breast cancer surgery. Cancer Nurs. 2014 Nov-Dec;37(6):406-17. doi: 10.1097/NCC.0000000000000131. PMID 24633334
- [Background] Lagendijk M, van Egdom LSE, Richel C, van Leeuwen N, Verhoef C, Lingsma HF, Koppert LB. Patient reported outcome measures in breast cancer patients. Eur J Surg Oncol. 2018 Jul;44(7):963-968. doi: 10.1016/j.ejso.2018.03.009. Epub 2018 Mar 21. PMID 29678302
- [Background] LeBlanc M, Stineman M, DeMichele A, Stricker C, Mao JJ. Validation of QuickDASH outcome measure in breast cancer survivors for upper extremity disability. Arch Phys Med Rehabil. 2014 Mar;95(3):493-8. doi: 10.1016/j.apmr.2013.09.016. Epub 2013 Oct 2. PMID 24095658
- [Background] Lewis SJ. Finding my own voice through the breast cancer journey: humour, sadness and smurfs. J Med Radiat Sci. 2015 Mar;62(1):82-5. doi: 10.1002/jmrs.92. No abstract available. PMID 26229671
- [Background] Lockefeer JP, De Vries J. What is the relationship between trait anxiety and depressive symptoms, fatigue, and low sleep quality following breast cancer surgery? Psychooncology. 2013 May;22(5):1127-33. doi: 10.1002/pon.3115. Epub 2012 Jun 13. PMID 22692984
- [Background] Machin, D., Campbell, M., Fayers, P., & Pinol, A. (1997). Sample size tables for clinical studies (2nd ed.). Oxford: Blackwell Science
- [Background] Madore S, Kilbourn K, Valverde P, Borrayo E, Raich P. Feasibility of a psychosocial and patient navigation intervention to improve access to treatment among underserved breast cancer patients. Support Care Cancer. 2014 Aug;22(8):2085-93. doi: 10.1007/s00520-014-2176-5. Epub 2014 Mar 18. PMID 24639035
- [Background] Mansano-Schlosser TC, Ceolim MF, Valerio TD. Poor sleep quality, depression and hope before breast cancer surgery. Appl Nurs Res. 2017 Apr;34:7-11. doi: 10.1016/j.apnr.2016.11.010. Epub 2016 Nov 17. PMID 28342628
- [Background] Matthews H, Carroll N, Renshaw D, Turner A, Park A, Skillman J, McCarthy K, Grunfeld EA. Predictors of satisfaction and quality of life following post-mastectomy breast reconstruction. Psychooncology. 2017 Nov;26(11):1860-1865. doi: 10.1002/pon.4397. Epub 2017 Mar 6. PMID 28195672
- [Background] Matthews, J.N.S. (2006). Introduction to randomized controlled clinical trials. 2nd Ed., Boca Raton, FL: Chapman & Hall/CRC.
- [Background] Min YH, Lee JW, Shin YW, Jo MW, Sohn G, Lee JH, Lee G, Jung KH, Sung J, Ko BS, Yu JH, Kim HJ, Son BH, Ahn SH. Daily collection of self-reporting sleep disturbance data via a smartphone app in breast cancer patients receiving chemotherapy: a feasibility study. J Med Internet Res. 2014 May 23;16(5):e135. doi: 10.2196/jmir.3421. PMID 24860070
- [Background] Mitchell S, Gass J, Hanna M. How Well Informed Do Patients Feel about Their Breast Cancer Surgery Options? Findings from a Nationwide Survey of Women after Lumpectomy and/or Mastectomy. J Am Coll Surg. 2018 Feb;226(2):134-146.e3. doi: 10.1016/j.jamcollsurg.2017.10.022. Epub 2017 Dec 12. PMID 29246706
- [Background] Morrow, J. (2012). Abstract LB-56: My journey as a breast cancer survivor, from diagnosis to advocate. Cancer Research, 72(8 Supplement), LB-56-LB-56. doi:10.1158/1538-7445.AM2012-LB-56
- [Background] Munro, B. H. (2005). Statistical Methods for Health Care Research (5th ed.). United States of America: Lippincott Williams & Wilkins.
- [Background] Ng CG, Mohamed S, Kaur K, Sulaiman AH, Zainal NZ, Taib NA; MyBCC Study group. Perceived distress and its association with depression and anxiety in breast cancer patients. PLoS One. 2017 Mar 15;12(3):e0172975. doi: 10.1371/journal.pone.0172975. eCollection 2017. PMID 28296921
- [Background] Nguyen J, Popovic M, Chow E, Cella D, Beaumont JL, Chu D, DiGiovanni J, Lam H, Pulenzas N, Bottomley A. EORTC QLQ-BR23 and FACT-B for the assessment of quality of life in patients with breast cancer: a literature review. J Comp Eff Res. 2015 Mar;4(2):157-66. doi: 10.2217/cer.14.76. PMID 25825844
- [Background] O'Regan P, Landers M, Hegarty J. A theoretical framework to guide a study exploring cancer related fatigue. Appl Nurs Res. 2017 Oct;37:19-23. doi: 10.1016/j.apnr.2017.07.003. Epub 2017 Jul 21. No abstract available. PMID 28985915
- [Background] Polit, D. F., & Beck, C. T. (2008b). Nursing Research:Principles and Methods. (8th ed.). Philadelphia: Lippincott Williams & Wilkins.
- [Background] Radina ME, Armer JM, Stewart BR. Making self-care a priority for women at risk of breast cancer-related lymphedema. J Fam Nurs. 2014 May;20(2):226-49. doi: 10.1177/1074840714520716. Epub 2014 Jan 29. PMID 24476674
- [Background] Rajaram N, Lim ZY, Song CV, Kaur R, Mohd Taib NA, Muhamad M, Ong WL, Schouwenburg M, See MH, Teo SH, Saunders C, Yip CH. Patient-reported outcome measures among breast cancer survivors: A cross-sectional comparison between Malaysia and high-income countries. Psychooncology. 2019 Jan;28(1):147-153. doi: 10.1002/pon.4924. Epub 2018 Oct 30. PMID 30346074
- [Background] Saboonchi F, Petersson LM, Wennman-Larsen A, Alexanderson K, Brannstrom R, Vaez M. Changes in caseness of anxiety and depression in breast cancer patients during the first year following surgery: patterns of transiency and severity of the distress response. Eur J Oncol Nurs. 2014 Dec;18(6):598-604. doi: 10.1016/j.ejon.2014.06.007. Epub 2014 Jul 2. PMID 24997517
- [Background] Saboonchi F, Wennman-Larsen A, Alexanderson K, Petersson LM. Examination of the construct validity of the Swedish version of Hospital Anxiety and Depression Scale in breast cancer patients. Qual Life Res. 2013 Dec;22(10):2849-56. doi: 10.1007/s11136-013-0407-8. Epub 2013 Apr 9. PMID 23568598
- [Background] Sandelowski M. What's in a name? Qualitative description revisited. Res Nurs Health. 2010 Feb;33(1):77-84. doi: 10.1002/nur.20362. PMID 20014004
- [Background] Schulz KF, Grimes DA. Allocation concealment in randomised trials: defending against deciphering. Lancet. 2002 Feb 16;359(9306):614-8. doi: 10.1016/S0140-6736(02)07750-4. PMID 11867132
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON
- [Background] Wallwiener M, Matthies L, Simoes E, Keilmann L, Hartkopf AD, Sokolov AN, Walter CB, Sickenberger N, Wallwiener S, Feisst M, Gass P, Fasching PA, Lux MP, Wallwiener D, Taran FA, Rom J, Schneeweiss A, Graf J, Brucker SY. Reliability of an e-PRO Tool of EORTC QLQ-C30 for Measurement of Health-Related Quality of Life in Patients With Breast Cancer: Prospective Randomized Trial. J Med Internet Res. 2017 Sep 14;19(9):e322. doi: 10.2196/jmir.8210. PMID 28912116
- [Background] Wang YJ, Boehmke M, Wu YW, Dickerson SS, Fisher N. Effects of a 6-week walking program on Taiwanese women newly diagnosed with early-stage breast cancer. Cancer Nurs. 2011 Mar-Apr;34(2):E1-13. doi: 10.1097/NCC.0b013e3181e4588d. PMID 20697267
- [Background] Wellisch, D., & Yarema, V. (2016). Coping together, side by side: Enriching mother-daughter communication across the breast cancer journey. written by carla L.fisher. hampton press inc., new york, NY, 2014. 242 pp. price: $29.95 (US), ₤17.01 (UK). ISBN: 978-1612891415 (paperbound). Psycho-Oncology, 25(6), 744-744. doi:10.1002/pon.4122
- [Background] Wen KY, Fang CY, Ma GX. Breast cancer experience and survivorship among Asian Americans: a systematic review. J Cancer Surviv. 2014 Mar;8(1):94-107. doi: 10.1007/s11764-013-0320-8. Epub 2013 Nov 9. PMID 24214498
- [Background] Wren AA, Shelby RA, Soo MS, Huysmans Z, Jarosz JA, Keefe FJ. Preliminary efficacy of a lovingkindness meditation intervention for patients undergoing biopsy and breast cancer surgery: A randomized controlled pilot study. Support Care Cancer. 2019 Sep;27(9):3583-3592. doi: 10.1007/s00520-019-4657-z. Epub 2019 Jan 31. PMID 30706142
- [Background] Xia J, Tang Z, Wu P, Wang J, Yu J. Use of item response theory to develop a shortened version of the EORTC QLQ-BR23 scales. Sci Rep. 2019 Feb 11;9(1):1764. doi: 10.1038/s41598-018-37965-x. PMID 30741988
- [Background] Yi, X., Gao, D., Gao, Z., Wang, Y. "., Yu, Z., Meng, K., . . . Yan, J. (2017). Smartphone application to home-based exercise on psychological wellbeing and physical functioning for breast cancer survivors: 3169 board #74 june 2 2. Medicine & Science in Sports & Exercise, 49, 896. doi:10.1249/01.mss.0000519433.34308.b7
- [Background] Zhao W. Selection bias, allocation concealment and randomization design in clinical trials. Contemp Clin Trials. 2013 Sep;36(1):263-5. doi: 10.1016/j.cct.2013.07.005. Epub 2013 Jul 19. No abstract available. PMID 23871796
- [Background] Zhu J, Ebert L, Liu X, Chan SW. A mobile application of breast cancer e-support program versus routine Care in the treatment of Chinese women with breast cancer undergoing chemotherapy: study protocol for a randomized controlled trial. BMC Cancer. 2017 Apr 26;17(1):291. doi: 10.1186/s12885-017-3276-7. PMID 28446141
- [Result] Alesia, A. (2015). Easing the breast cancer journey. Business People, 28(11), 20.
- [Derived] Pang Y, He H, Ng RP, Lee NKL, Htein MMW, Zhao XX, Li YH, Chan EJ, Zhu L, Liu GY, Pikkarainen M, Lim SH. Effectiveness of an Innovative Mobile-Based Perioperative Care Program for Women Undergoing Breast Cancer Surgery (iCareBreast): Randomized Controlled Trial. J Med Internet Res. 2025 Apr 21;27:e71684. doi: 10.2196/71684. PMID 40258266
- See also: Cancer Statistics — https://www.nccs.com.sg/patient-care/cancer-types/cancer-statistics
- See also: Khalik, S. (2017, June 20). Breast, prostate cancers rising sharply in Singapore. — https://www.straitstimes.com/singapore/health/breast-prostate-cancers-rising-sharply-in-spore
- See also: National Cancer Centre Singapore. (2017). Obesity and Breast Cancer. — https://www.nccs.com.sg/news/medical-news-singhealth/obesity-and-breast-cancer